CLINICAL TRIAL: NCT00149383
Title: A Randomized, Double-blind, Placebo-controlled Trial of Rosiglitazone as Adjunctive Therapy for P.Falciparum Infection
Brief Title: Safety and Efficacy Study of Adjunctive Rosiglitazone in the Treatment of Uncomplicated Falciparum Malaria
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: McLaughlin-Rotman Center for Global Health, University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 033-2004
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-04

CONDITIONS: Falciparum Malaria
Keywords: randomized controlled trial; malaria; Plasmodium falciparum; thiazolidinediones; rosiglitazone; atovaquone-proguanil
MeSH Terms: conditions — Malaria, Falciparum; Malaria | interventions — Rosiglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo
- 1 (Experimental)
  Interventions: Drug: Rosiglitazone

INTERVENTIONS:
Drug: Rosiglitazone
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
The purpose of this study is to examine the safety, tolerability, and efficacy of adjunctive rosiglitazone in the treatment of uncomplicated P.falciparum malaria.

DETAILED DESCRIPTION:
Study Rationale: Evidence suggests that if PPAR-RXR agonists (such as rosiglitazone) are used as adjunctive therapy in P. falciparum malaria infections they may increase phagocytic clearance of P. falciparum malaria, modulate deleterious inflammatory responses and decrease sequestration of malaria parasites in vital organs. They may therefore represent a novel immunomodulatory treatment approach for P. falciparum malaria.

Study Objectives: 1) To examine the in vivo effect of rosiglitazone on the rapidity of clearance of P. falciparum parasitemia and fever in patients with non-severe P. falciparum infections 2) To assess the safety and tolerability of adjunctive rosiglitazone treatment in non-severe cases of P. falciparum infection.

Primary Outcomes: Time to clearance of P. falciparum parasitemia

Study Design: Randomized double blind placebo-controlled trial.

Intervention: Standard antimalarial treatment (atovaquone/proguanil) to all patients combined with adjuvant rosiglitazone treatment (8mg per day) or placebo.

Setting: Hospital for Tropical Diseases at Mahidol University, Thailand.

Participants: 140 patients with non-severe P. falciparum infection.

Follow-up: 28 days

ELIGIBILITY:
Inclusion Criteria:

* Microscopically confirmed P.falciparum infection
* Age >18 years
* Able to tolerate oral therapy
* Able to give informed consent

Exclusion Criteria:

* Fulfillment of WHO criteria for severe/cerebral malaria
* Prior treatment with any thiazolidinedione
* Allergy to rosiglitazone
* History of diabetes mellitus
* History of severe/decompensated liver disease
* ALT level >2.5 times normal
* Current treatment for congestive heart failure
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2004-12; Primary Completion 2005-11 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Time to clearance (in hours) of parasitemia from blood is recorded | 5 days

SECONDARY OUTCOMES:
Time to resolution of fever (in hours) | 5 days
AST/ALT levels (U/L) | 2 days
Capillary blood glucose (mmol/L) | 2 days
Need for ICU admission | 5 days
Tolerability of study drug/placebo as assessed by patient log | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Kevin C Kain, MD, FRCPC, Principal Investigator — Faculty of Medicine, University of Toronto; McLaughlin-Rotman Center for Global Health, Toronto
Locations (1):
- Faculty of Tropical Medicine, Mahidol University, Bangkok, Thailand

REFERENCES:
- [Background] Suh KN, Kain KC, Keystone JS. Malaria. CMAJ. 2004 May 25;170(11):1693-702. doi: 10.1503/cmaj.1030418. PMID 15159369
- [Background] Patel SN, Serghides L, Smith TG, Febbraio M, Silverstein RL, Kurtz TW, Pravenec M, Kain KC. CD36 mediates the phagocytosis of Plasmodium falciparum-infected erythrocytes by rodent macrophages. J Infect Dis. 2004 Jan 15;189(2):204-13. doi: 10.1086/380764. Epub 2004 Jan 9. PMID 14722884
- [Background] Serghides L, Smith TG, Patel SN, Kain KC. CD36 and malaria: friends or foes? Trends Parasitol. 2003 Oct;19(10):461-9. doi: 10.1016/j.pt.2003.08.006. No abstract available. PMID 14519584
- [Background] Smith TG, Ayi K, Serghides L, Mcallister CD, Kain KC. Innate immunity to malaria caused by Plasmodium falciparum. Clin Invest Med. 2002 Dec;25(6):262-72. PMID 12516999
- [Background] Smith TG, Serghides L, Patel SN, Febbraio M, Silverstein RL, Kain KC. CD36-mediated nonopsonic phagocytosis of erythrocytes infected with stage I and IIA gametocytes of Plasmodium falciparum. Infect Immun. 2003 Jan;71(1):393-400. doi: 10.1128/IAI.71.1.393-400.2003. PMID 12496189
- [Background] Serghides L, Kain KC. Mechanism of protection induced by vitamin A in falciparum malaria. Lancet. 2002 Apr 20;359(9315):1404-6. doi: 10.1016/S0140-6736(02)08360-5. PMID 11978340
- [Background] Serghides L, Kain KC. Peroxisome proliferator-activated receptor gamma-retinoid X receptor agonists increase CD36-dependent phagocytosis of Plasmodium falciparum-parasitized erythrocytes and decrease malaria-induced TNF-alpha secretion by monocytes/macrophages. J Immunol. 2001 Jun 1;166(11):6742-8. doi: 10.4049/jimmunol.166.11.6742. PMID 11359831
- [Background] McGilvray ID, Serghides L, Kapus A, Rotstein OD, Kain KC. Nonopsonic monocyte/macrophage phagocytosis of Plasmodium falciparum-parasitized erythrocytes: a role for CD36 in malarial clearance. Blood. 2000 Nov 1;96(9):3231-40. PMID 11050008
- [Background] Serghides L, Crandall I, Hull E, Kain KC. The Plasmodium falciparum-CD36 interaction is modified by a single amino acid substitution in CD36. Blood. 1998 Sep 1;92(5):1814-9. PMID 9716613
- [Background] Urquhart AD. Putative pathophysiological interactions of cytokines and phagocytic cells in severe human falciparum malaria. Clin Infect Dis. 1994 Jul;19(1):117-31. doi: 10.1093/clinids/19.1.117. PMID 7948512
- [Background] Ockenhouse CF, Ho M, Tandon NN, Van Seventer GA, Shaw S, White NJ, Jamieson GA, Chulay JD, Webster HK. Molecular basis of sequestration in severe and uncomplicated Plasmodium falciparum malaria: differential adhesion of infected erythrocytes to CD36 and ICAM-1. J Infect Dis. 1991 Jul;164(1):163-9. doi: 10.1093/infdis/164.1.163. PMID 1711552
- [Background] Ockenhouse CF, Chulay JD. Plasmodium falciparum sequestration: OKM5 antigen (CD36) mediates cytoadherence of parasitized erythrocytes to a myelomonocytic cell line. J Infect Dis. 1988 Mar;157(3):584-8. doi: 10.1093/infdis/157.3.584. No abstract available. PMID 2449507
- [Background] Oquendo P, Hundt E, Lawler J, Seed B. CD36 directly mediates cytoadherence of Plasmodium falciparum parasitized erythrocytes. Cell. 1989 Jul 14;58(1):95-101. doi: 10.1016/0092-8674(89)90406-6. PMID 2473841
- [Background] Day NP, Hien TT, Schollaardt T, Loc PP, Chuong LV, Chau TT, Mai NT, Phu NH, Sinh DX, White NJ, Ho M. The prognostic and pathophysiologic role of pro- and antiinflammatory cytokines in severe malaria. J Infect Dis. 1999 Oct;180(4):1288-97. doi: 10.1086/315016. PMID 10479160
- [Background] Kwiatkowski D, Hill AV, Sambou I, Twumasi P, Castracane J, Manogue KR, Cerami A, Brewster DR, Greenwood BM. TNF concentration in fatal cerebral, non-fatal cerebral, and uncomplicated Plasmodium falciparum malaria. Lancet. 1990 Nov 17;336(8725):1201-4. doi: 10.1016/0140-6736(90)92827-5. PMID 1978068
- [Background] Brown H, Turner G, Rogerson S, Tembo M, Mwenechanya J, Molyneux M, Taylor T. Cytokine expression in the brain in human cerebral malaria. J Infect Dis. 1999 Nov;180(5):1742-6. doi: 10.1086/315078. PMID 10515846
- [Background] Aitman TJ, Cooper LD, Norsworthy PJ, Wahid FN, Gray JK, Curtis BR, McKeigue PM, Kwiatkowski D, Greenwood BM, Snow RW, Hill AV, Scott J. Malaria susceptibility and CD36 mutation. Nature. 2000 Jun 29;405(6790):1015-6. doi: 10.1038/35016636. No abstract available. PMID 10890433
- [Background] Omi K, Ohashi J, Naka I, Patarapotikul J, Hananantachai H, Looareesuwan S, Tokunaga K. Polymorphisms of CD36 in Thai malaria patients. Southeast Asian J Trop Med Public Health. 2002;33 Suppl 3:1-4. PMID 12971464
- [Background] Shankar AH, Genton B, Semba RD, Baisor M, Paino J, Tamja S, Adiguma T, Wu L, Rare L, Tielsch JM, Alpers MP, West KP Jr. Effect of vitamin A supplementation on morbidity due to Plasmodium falciparum in young children in Papua New Guinea: a randomised trial. Lancet. 1999 Jul 17;354(9174):203-9. doi: 10.1016/S0140-6736(98)08293-2. PMID 10421302
- [Background] Schoonjans K, Auwerx J. Thiazolidinediones: an update. Lancet. 2000 Mar 18;355(9208):1008-10. doi: 10.1016/S0140-6736(00)90002-3. PMID 10768450
- [Derived] Boggild AK, Krudsood S, Patel SN, Serghides L, Tangpukdee N, Katz K, Wilairatana P, Liles WC, Looareesuwan S, Kain KC. Use of peroxisome proliferator-activated receptor gamma agonists as adjunctive treatment for Plasmodium falciparum malaria: a randomized, double-blind, placebo-controlled trial. Clin Infect Dis. 2009 Sep 15;49(6):841-9. doi: 10.1086/605431. PMID 19673614
- See also: Mahidol University, Faculty of Tropical Medicine — http://www.tm.mahidol.ac.th